CLINICAL TRIAL: NCT02314689
Title: A Dose Escalation Study of Intravenous L-citrulline in Steady-state Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suvankar Majumdar (Other)
Responsible Party: Sponsor-Investigator, Suvankar Majumdar, Associate Professor, University of Mississippi Medical Center
Organization: University of Mississippi Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCD-124700.
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Citrulline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV citrulline (Experimental): IV citrulline 20 mg/kg bolus with dose escalation of 10 mg/kg to target citrulline concentration of 100 µmol/L with a maximum dose of 60 mg/kg.
  Interventions: Drug: Intravenous (IV) citrulline

INTERVENTIONS:
Drug: Intravenous (IV) citrulline

SUMMARY:
The purpose of this study is to assess the maximum tolerated dose, safety and pharmacokinetics of an investigational drug, intravenous (IV) citrulline, in subjects in steady-state sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease genotypes (HbSS, HbS/β° thalassemia, HbS/β+thalassemia, HbSC)

Exclusion Criteria:

* Presence of any acute illness defined by fever >100.4° F within the past 48 hours
* Presence of sickle cell pain crisis defined by the presence of pain requiring oral or parental opioid therapy.
* Presence of acute chest syndrome or presence of any other complication related to sickle cell disease requiring hospitalization such as splenic sequestration, hepatic sequestration, stroke, avascular necrosis of the hip/shoulder, acute priapism, and patients with diabetes etc.
* Severe anemia (hemoglobin < 5g/dL)
* History of red blood cell transfusion within the last 14 days
* Systemic steroid therapy within the last 48 hours
* Pregnant (as confirmed by a negative urine pregnancy test) or lactating female
* Alanine/aspartate transferase >2x upper limit of normal laboratory range for age.
* Elevated serum creatinine >1.5mg/dL
* Patients with an inability to give consent will be excluded
* Medications that are known to be contra-indicated with use of L-citrulline (concurrent use of hydroxyurea will be allowed).
* History of diabetes due to risk of electrolyte imbalance

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Barr FE, Tirona RG, Taylor MB, Rice G, Arnold J, Cunningham G, Smith HA, Campbell A, Canter JA, Christian KG, Drinkwater DC, Scholl F, Kavanaugh-McHugh A, Summar ML. Pharmacokinetics and safety of intravenously administered citrulline in children undergoing congenital heart surgery: potential therapy for postoperative pulmonary hypertension. J Thorac Cardiovasc Surg. 2007 Aug;134(2):319-26. doi: 10.1016/j.jtcvs.2007.02.043. PMID 17662768

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous (IV) Citrulline: Intravenous (IV) citrulline 20 mg/kg bolus with dose escalation of 10 mg/kg to target citrulline concentration of 100 µmol/L with a maximum dose of 60 mg/kg.
Period: Overall Study
Arm/Group | Intravenous (IV) Citrulline
Started | 4
Completed | 4 (Target citrulline level reached with first 4 subjects enrolled at initial IV citrulline of 20 mg/kg)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intravenous (IV) Citrulline
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 22.8 [21 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Adverse Event According to NCI Criteria
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- IV Citrulline: IV citrulline 20 mg/kg bolus with dose escalation of 10 mg/kg to target citrulline concentration of 100 µmol/L with a maximum dose of 60 mg/kg.
  Intravenous (IV) citrulline
Arm/Group | IV Citrulline
Number analyzed (Participants) | 4
participants | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Intravenous (IV) Citrulline
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous (IV) Citrulline (N=4)
Greater than 20% drop in blood pressure (Vascular disorders) | 1 (1) — 1 out of the 4 patients dropped the DBS greater than 20% from baseline but maintained normal systolic BP, heart rate and other vital signs. Participant did not require any intervention. Case was reviewed by the DSMB and deemed a grade 1 adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes